CLINICAL TRIAL: NCT00717977
Title: A Study to Assess Continuous Glucose Sensor Profiles in Healthy Non-Diabetic Subjects
Brief Title: Continuous Glucose Sensor Profiles in Non-Diabetic Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: JDRF Artificial Pancreas Project (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2008-2403
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects Without Type 1 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Continuous glucose monitor — Daily use of a continuous glucose monitor for 3-7 days
  Other Names: Abbott FreeStyle Navigator; DexCom SEVEN; Medtronic Guardian Clinical

SUMMARY:
The Juvenile Diabetes Research Foundation (JDRF) Glucose Sensor Study group is carrying out a large, randomized clinical trial to assess the efficacy, safety and cost-effectiveness of use of real-time continuous glucose monitors (RT-CGM) as an adjunct to standard meter plasma glucose testing. Although the primary outcome in the >= 7.0% cohort is differences in HbA1c levels, important secondary outcomes are differences in the percent of glucose sensor values either above or below the target glucose range of 70-180 mg/dl and differences in glucose variability. Prevention of biochemical hypoglycemia is a particularly important outcome in the low HbA1c cohort. Since CGM systems measure interstitial rather than plasma glucose and CGM values differ from simultaneous plasma glucose values by up to 18%, it would be extremely useful for comparative purposes to establish a reference range of sensor values in healthy, non-diabetic control subjects for this study and other future investigations. The objective of this protocol is to establish such reference sensor glucose ranges in each of the 3 devices being utilized in the JDRF study.

DETAILED DESCRIPTION:
1. After initial eligibility is determined, informed consent and assent are obtained from the parent/guardian and subject.
2. Subjects will have the following tests performed:

   * Hemoglobin A1c (using the DCA2000 or equivalent device)
   * Oral glucose tolerance test to obtain fasting and 2 hour plasma glucose levels
   * Anti-GAD, anti-IA2 and anti-insulin antibodies

     * Subjects with an HbA1c >6.0% and/or fasting glucose levels >100 and/or 2 hour glucose levels >140 will be discontinued from the study.
3. Subjects with normal A1c and glucose levels will be provided with an RT-CGM and home glucose meter (HGM)
4. An RT-CGM sensor will be inserted and initiated by study personnel.
5. Subjects who would like to wear 2 sensors will be given 2 of the same type of RT-CGM.
6. Subjects will be instructed to wear the sensor for 3-7 days (depending on the type of device) and measure the blood glucose on the HGM as needed to calibrate the sensor.
7. Subjects will return to the clinical center after the 3-7 days of sensor wear to return the RT-CGM and HGM.

   * If the subject has less than 48 hours of sensor data he or she will be asked to wear another sensor and return 3-7 days later.

ELIGIBILITY:
Inclusion Criteria:

* Age > 8 years
* Body mass index (BMI) between the 10th to 90th percentile for age and sex (based on CDC, 2000 nomogram) and < 28 kg body weight/meter in adult subjects
* No significant chronic illness or taking any acute or chronic medications that might affect glucose metabolism.

Exclusion Criteria:

* History of diabetes or positive islet cell antibody testing

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, M.D., Ph.D., Study Director — Jaeb Center for Health Research; Lori Laffel, M.D., Study Chair — Joslin Diabetes Center Pediatric Section; William Tamborlane, M.D., Study Chair — Yale University
Locations (10):
- United States (10):
  - Kaiser Permanente, San Diego, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Children's Hospital of Iowa, Iowa City, Iowa
  - Joslin Diabetes Center - Adults, Boston, Massachusetts
  - Joslin Diabetes Center - Children, Boston, Massachusetts
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Fox LA, Beck RW, Xing D. Variation of interstitial glucose measurements assessed by continuous glucose monitors in healthy, nondiabetic individuals. Diabetes Care. 2010 Jun;33(6):1297-9. doi: 10.2337/dc09-1971. Epub 2010 Mar 9. PMID 20215454
- [Derived] Shah VN, Vigers T, Pyle L, Calhoun P, Bergenstal RM. Discordance Between Glucose Management Indicator and Glycated Hemoglobin in People Without Diabetes. Diabetes Technol Ther. 2023 May;25(5):324-328. doi: 10.1089/dia.2022.0544. Epub 2023 Mar 3. PMID 36790875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 adult and pediatric diabetes centers, after approval by their institutional review boards. Subjects were healthy adults, adolescents, and children who were clinic staff, friends, relatives of clinic staff, or relatives or acquaintances of an individual with type 1 diabetes.
Groups:
- All Non-Diabetic Subjects: Subjects were healthy adults, adolescents, and children who were clinic staff, friends, relatives of clinic staff, or relatives or acquaintances of an indiviual with type 1 diabetes.
Period: Overall Study
Arm/Group | All Non-Diabetic Subjects
Started | 74
Completed | 74
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Age, Customized [Number; unit: Participants]
  8-<15 years | 20
  15-<25 years | 17
  25-<45 years | 20
  >=45 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 23
Race/Ethnicity, Customized [Number; unit: Participant]
  Non-Hispanic, Caucasian | 55
  Hispanic | 13
  African American | 1
  Other Race/Ethnicities | 5
2-hour post-oral glucose tolerance test (OGTT) [Mean (Standard Deviation); unit: mg/dL] — Fasting blood glucose measurement taken 2 hours following the OGTT.
  mg/dL | 96 (22)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 86 (8)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent]
  All | 5.3 (0.3)
  8-<15 years | 5.3 (0.2)
  15-<25 years | 5.2 (0.2)
  25-<45 years | 5.2 (0.3)
  >=45 years | 5.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Sensor Glucose by Age Group
Description: Mean glucose value was calculated for every hour of the 24 hours of the day. This measure is the average over all 24 hours.
Time Frame: 48-72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 98 (10)
  8-<15 years | 103 (11)
  15-<25 years | 97 (7)
  25-<45 years | 96 (12)
  >=45 years | 95 (7)
Statistical Analysis 1: Comparison: All Non-Diabetic Subjects; The associations of mean sensor glucose and glucose variability measures with age were assessed using least-squares regression models adjusting for device type; Test type: Superiority or Other; p = 0.009, Regression, Linear — Adjusted for CGM device type. Age was analyzed as continuous

2. Primary Outcome: Daytime (6:00 a.m. - Midnight) Mean Sensor Glucose by Age Group
Description: Mean glucose value was calculated for every hour of the 24 hours of the day. This measure is the average from 6 a.m. to midnight.
Time Frame: 48-72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 99 (10)
  8-<15 years | 103 (10)
  15-<25 years | 98 (7)
  25-<45 years | 97 (12)
  >=45 years | 97 (6)
Statistical Analysis 1: Comparison: All Non-Diabetic Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.04, Regression, Linear — Adjusted for CGM device type. Age was analyzed as continuous

3. Primary Outcome: Nighttime (Midnight - 6:00 a.m.) Mean Sensor Glucose by Age Group
Description: Mean glucose value was calculated for every hour of the 24 hours of the day. This measure is the average from midnight to 6 a.m.
Time Frame: 48-72 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 95 (13)
  8-<15 years | 101 (15)
  15-<25 years | 97 (11)
  25-<45 years | 91 (12)
  >=45 years | 89 (11)
Statistical Analysis 1: Comparison: All Non-Diabetic Subjects; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Linear — Adjusted for device type. Age was analyzed as continuous

4. Primary Outcome: Peak Daytime Sensor Glucose Value by Age Group
Description: The calculation of peak and nadir glucose was restricted to days with >=12 hours and nights with >=4 hours of sensor glucose data.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 131 [121 to 140]
  8-<15 years | 134 [128 to 145]
  15-<25 years | 135 [119 to 144]
  25-<45 years | 125 [118 to 134]
  >=45 years | 128 [122 to 134]

5. Primary Outcome: Peak Nightime Sensor Glucose Value by Age Group
Description: as for outcome 4
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 109 [99 to 118]
  8-<15 years | 111 [108 to 120]
  15-<25 years | 111 [106 to 118]
  25-<45 years | 104 [95 to 111]
  >=45 years | 103 [97 to 113]

6. Primary Outcome: Daytime Nadir Sensor Glucose Value by Age Group
Description: The calculation of peak and nadir glucose was restricted to days with >=12 hours and nights with >=4 hours of sensor glucose data. The daytime nadir reflects the lowest point on the sensor glucose curve registered among daytime values.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 73 [68 to 82]
  8-<15 Years | 74 [68 to 86]
  15-<25 Years | 71 [67 to 77]
  25-<45 Years | 75 [67 to 82]
  >=45 Years | 79 [68 to 84]

7. Primary Outcome: Nighttime Nadir Sensor Glucose Value by Age Group
Description: The calculation of peak and nadir glucose was restricted to days with >=12 hours and nights with >=4 hours of sensor glucose data. The nighttime nadir reflects the lowest point on the sensor glucose curve registered among nighttime values.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 80 [73 to 89]
  5-<15 Years | 84 [78 to 91]
  15-<25 Years | 80 [76 to 93]
  25-<45 Years | 77 [67 to 88]
  >=45 Years | 78 [78 to 86]

8. Primary Outcome: Percentage of Sensor Glucose Levels Between 71-120 mg/dL by Age Group
Description: The Percentage Sensor Glucose Levels between 71-120 mg/dL was calculated for each subject. The median and quartiles over all subjects were reported here.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 91.0 [79 to 94]
  8-<15 Years | 85.1 [79 to 92]
  15-<25 Years | 87.9 [76 to 96]
  25-<45 Years | 91.4 [78 to 94]
  >=45 Years | 93.7 [88 to 95]

9. Primary Outcome: Percentage of Sensor Glucose Levels 71-120 mg/dL by Time of Day
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 90.4 [80 to 95]
  Nightime (midnight-6am) | 90.3 [76 to 98]

10. Primary Outcome: Distribution of Sensor Glucose Levels <=70 mg/dL by Age Group
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 1.7 [0.0 to 7.2]
  8-<15 Years | 1.8 [0.0 to 4.3]
  15-<25 Years | 0.6 [0.0 to 8.1]
  25-<45 Years | 2.9 [0.0 to 8.1]
  >=45 Years | 1.6 [0.0 to 6.3]

11. Primary Outcome: Percentage of Sensor Glucose Levels <=70 mg/dl by Time of Day
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 1.1 [0.0 to 5.1]
  Nighttime (midnight-6am) | 2.2 [0.0 to 12]

12. Primary Outcome: Percentage of Sensor Glucose Levels <=60 mg/dL by Age Group
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 0.2 [0.0 to 1.7]
  8-<15 Years | 0.2 [0.0 to 1.8]
  15-<25 Years | 0.0 [0.0 to 3.1]
  25-<45 Years | 0.2 [0.0 to 1.3]
  >=45 Years | 0.1 [0.0 to 1.3]

13. Primary Outcome: Percentage of Sensor Glucose Levels <=60 mg/dl by Time of Day
Description: The Percentage of Sensor Glucose Levels <=60 mg/dl was calculated for each subject separately for the daytime and nighttime period. The median and quartiles over all subjects were reported.
  Here the data is different with data analyzed by age group, which is a subgroup analysis on 'percentage of sensor glucose levels <=60mg/dL' for all 24 hours.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 0.0 [0.0 to 1.2]
  Nighttime (midnight-6am) | 0.0 [0.0 to 1.3]

14. Primary Outcome: Percentage of Sensor Glucose Levels >120 mg/dL by Age Group
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 5.6 [2.2 to 9.3]
  8-<15 Years | 8.2 [5.6 to 16]
  15-<25 Years | 8.3 [3.1 to 13]
  25-<45 Years | 4.2 [1.8 to 7.1]
  >=45 Years | 4.4 [1.2 to 5.8]

15. Primary Outcome: Percentage of Sensor Glucose Levels >120 mg/dl by Time of Day
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 5.9 [2.4 to 11]
  Nighttime (midnight-6am) | 1.1 [0.0 to 11]

16. Primary Outcome: Percentage of Sensor Glucose Levels >140 mg/dL by Age Group
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 0.4 [0.0 to 1.7]
  5-<15 Years | 1.3 [0.3 to 3.7]
  15-<25 Years | 0.3 [0.0 to 1.5]
  25-<45 Years | 0.3 [0.0 to 1.9]
  >=45 Years | 0.0 [0.0 to 1.0]

17. Primary Outcome: Percentage of Sensor Glucose Levels >140 mg/dl by Time of Day
Description: The Percentage of Sensor Glucose Levels >140 mg/dl was calculated for each subject separately for the daytime and nighttime period. The median and quartiles over all subjects were reported.
  Here the data is different with data analyzed by age group, which is a subgroup analysis on 'percentage of sensor glucose levels >140 mg/dl' for all 24 hours.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 0.5 [0.0 to 2.3]
  Nighttime (midnight-6am) | 0.0 [0.0 to 0.0]

18. Primary Outcome: Glucose Variability Measure- Standard Deviation by Age Group
Description: Here, 'Standard Deviation' is a measure of glucose variability. This measure was calculated by taking the SD of all glucose values for each subject. Each subject has a SD value. The median and quartiles of this measure over all subjects were reported.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 13.7 [11.4 to 18.0]
  8-<15 Years | 16.4 [13.2 to 19.1]
  15-<25 Years | 13.7 [11.1 to 19.9]
  25-<45 Years | 12.6 [12.1 to 16.5]
  >=45 Years | 12.4 [10.0 to 15.9]

19. Primary Outcome: Glucose Variability Measure- Standard Deviation by Time of Day
Description: as for outcome 18
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  Daytime (6am-midnight) | 13.5 [11.3 to 17.8]
  Nighttime (midnight-6am) | 10.9 [8.2 to 16.8]

20. Primary Outcome: Glucose Variability Measure- Absolute Rate of Change by Age Group
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL/min
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL/min
  All | 0.34 [0.30 to 0.41]
  8-<15 Years | 0.36 [0.36 to 0.46]
  15-<25 Years | 0.34 [0.30 to 0.39]
  25-<45 Years | 0.32 [0.28 to 0.37]
  >=45 Years | 0.33 [0.24 to 0.41]

21. Primary Outcome: Glucose Variability Measure- Absolute Rate of Change by Time of Day
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL/min
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL/min
  Daytime (6am-midnight) | 0.37 [0.32 to 0.43]
  Nighttime (midnight-6am) | 0.26 [0.18 to 0.35]

22. Primary Outcome: Glucose Variability Measure- Coefficient of Variation by Age Group
Description: The Coefficient of Variation is calculated by dividing the standard deviation by the mean glucose. Each subject received a SD value. The median and quartiles of this measure over all subjects were reported.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  All | 14 [12 to 19]
  8-<15 Years | 16 [13 to 19]
  15-<25 Years | 14 [12 to 21]
  25-<45 Years | 14 [13 to 17]
  >=45 Years | 13 [10 to 16]

23. Primary Outcome: Glucose Variability Measure- Coefficient of Variation by Time of Day
Description: as for outcome 22
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
Percent
  Daytime (6am-midnight) | 14 [12 to 18]
  Nighttime (midnight-6am) | 12 [9 to 19]

24. Primary Outcome: Glucose Variability Measure: Mean Amplitude of Glycemic Excursions by Age Group
Description: The Mean Amplitude of Glycemic Excursions also known as MAGE depicts the upward and downward acute glucose fluctuations seen in the sensor data.
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  All | 27.7 [23.1 to 33.1]
  8-<15 Years | 28.1 [23.9 to 33.2]
  15-<25 Years | 28.3 [25.1 to 33.1]
  25-<45 Years | 25.6 [22.8 to 31.4]
  >=45 Years | 26.9 [21.4 to 34.1]

25. Primary Outcome: Glucose Variability Measure: Amplitude of Glycemic Excursions by Time of Day
Description: as for outcome 24
Time Frame: 48-72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | All Non-Diabetic Subjects
Number analyzed (Participants) | 74
mg/dL
  Daytime (6am-midnight) | 28.0 [23.8 to 31.9]
  Nighttime (midnight-6am) | 15.8 [12.3 to 20.3]

ADVERSE EVENTS:
Arm/Group | All Non-Diabetic Subjects
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less